CLINICAL TRIAL: NCT07232498
Title: Early Doppler-Assisted Mobilization in Adults After Acute Ischemic Stroke - a Randomized Clinical Trial
Brief Title: Early Doppler-Assisted Mobilization in Adults After Acute Ischemic Stroke
Acronym: DOP-MOBILIZE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Collaborators: Unidade Local de Saúde São João (Other Government); Unidade Local de Saúde Santa Maria (Other Government)
Responsible Party: Principal Investigator, João Sargento Freitas, Principal Investigator, MD, PhD, Stroke Unit Coordinator, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 197/24 CE
Record Dates: First submitted 2025-09-16; First posted 2025-11-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Arterial Ischemic Stroke
Keywords: Arterial Ischemic Stroke; Early mobilization; mRS; Transcranial doppler ultrasound; Neurology; Hemodynamics
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doppler-guided early mobilization (Experimental): Patients with ischemic stroke will be mobilized based on the results of carotid and transcranial Doppler ultrasound examinations. If significant hemodynamic alterations are identified, such as stenosis ≥70% or intracranial occlusions, mobilization will be gradually introduced up to the 5th-7th day post-event. In the absence of such alterations, mobilization will begin immediately, with out-of-bed transfer to a chair within 48 hours and gait training, if clinically feasible.
  Interventions: Procedure: Doppler-guided early mobilization
- Standard Care Mobilization - Control Group (No Intervention): Patients with ischemic stroke are mobilized according to standard clinical practice, without considering hemodynamic assessment results from Doppler ultrasound. Mobilization is introduced gradually, guided by the patient's clinical tolerance.

INTERVENTIONS:
Procedure: Doppler-guided early mobilization — Individualized early mobilization after ischemic stroke, guided by hemodynamic assessment using carotid and transcranial Doppler ultrasound. The type and timing of mobilization are adjusted according to the presence of significant hemodynamic alterations.
  Arms: Doppler-guided early mobilization

SUMMARY:
Post-stroke mobilization remains a subject of ongoing debate. While early mobilization-particularly the first out-of-bed mobilization-has been associated with reduced systemic complications and earlier rehabilitation, it also carries potential risks, such as neurological deterioration in the presence of hemodynamic instability.

In this study, the primary aim is to investigate whether early mobilization, guided by hemodynamic evaluation after acute ischemic stroke offers superior outcomes compared to standard clinical care.

DETAILED DESCRIPTION:
Cerebrovascular diseases are the leading cause of death in Portugal and one of the most significant contributors to morbidity and disability.

Early mobilization after stroke is debated due to its potential benefits-such as fewer systemic complications and faster rehabilitation-and risks, particularly in patients with hemodynamic instability.

International guidelines support for early mobilization tailored to the patient's neurological status; however, the scientific evidence remains limited, resulting in heterogeneous practices across institutions.

Previous studies have highlighted the insufficient consideration of hemodynamic status when determining the timing of initial mobilization.

This study is a phase 3, pragmatic, prospective, multicenter randomized controlled trial with blinded outcome assessment (PROBE design: Prospective, Randomized, Open-label, Blinded Outcome Assessment), with an anticipated total duration of 36 months.

The study will be conducted in the Neurology Departments of the participating hospital centers and aims to: (1) evaluate the superiority of early mobilization guided by hemodynamic assessment following acute ischemic stroke, compared to standard clinical practice; (2) assess neurological deficits, quality of life, and cognitive function at three months, as well as hospital length of stay, blood pressure profile evolution, patient-reported outcome measures (PROMs), and employability; (3) compare adverse events between patients undergoing Doppler-guided early mobilization and those in the control group, including hospital-acquired infections, neurological deterioration, hemorrhagic transformation, and mortality.

Patients randomized to the intervention group will be mobilized according to carotid and transcranial Doppler ultrasound findings. In the presence of hemodynamic impairment, patients will undergo progressive mobilization, aiming to be out of bed by days 5 to 7 post-stroke, with gait training as neurologically feasible. In the absence of such findings, patients will begin mobilization immediately after the examination, with the goal of being out of bed and seated within 72 hours, including gait training when possible. Functional status at three months will be assessed using the modified Rankin Scale (mRS), which constitutes the study's primary endpoint.

All data collection procedures will follow formal and ethical research standards, ensuring that all informed participants voluntarily, anonymously, consent to take part in the study, with confidentiality maintained and no costs or harm to participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ischemic stroke aged 18 years or older;
* Ability to undergo carotid and transcranial Doppler ultrasound, as well as to mobilize within 48 hours;
* Informed consent obtained from the patient or legal representative.

Exclusion Criteria:

* Pre-existing disability with a modified Rankin Scale (mRS) score ≥ 4;
* Diagnosis of Transient Ischemic Attack (TIA);
* Severe hemodynamic instability, defined as:
* Systolic blood pressure < 100 mmHg or > 220 mmHg;
* Peripheral oxygen saturation < 92%;
* Heart rate < 40 or > 112 beats per minute;
* Body temperature > 38.5°C;
* Neurological deterioration with altered level of consciousness (defined as Glasgow Coma Scale < 10);
* Patients who underwent neurosurgical intervention within the past 30 days;
* Concomitant diagnosis of a rapidly progressive fatal disease (e.g., terminal-stage cancer);
* Requirement for continuous monitoring or continuous intravenous drug infusion;
* Acute deep vein thrombosis/pulmonary embolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Functional status at 3 months after ischemic stroke | 3 months post-stroke
  Functional status assessment at 3 months after ischemic stroke, using the modified Rankin Scale (mRS), analyzed on an ordinal scale (0-6), to measure the degree of dependence/functional impairment.
  Score ranges:
  0-no residual symptoms (better outcome);
  1. no significant disability;
  2. slight disability;
  3. moderate disability;
  4. moderately severe disability;
  5. severe disability;
  6. death (worse outcome).

SECONDARY OUTCOMES:
Neurological Assessment (NIHSS Scale) | Day 0, 48 hours, Day 7 and Month 3
  Neurological assessment on the 7th day after ischemic stroke, measured using the National Institutes of Health Stroke Scale score (NIHSS, from 0-42) to evaluate the severity of neurological deficits.
  Score ranges:
  0-4: Minor Stroke (better outcome); 5-15: Moderate Stroke; 16-20: Moderate to Severe Stroke; 21-42: Severe Stroke (worse outcome).
Development of hospital-acquired infections | Up to 7 days
  Incidence of infections acquired during hospitalization
Vital signs - Body temperature | Day 0, 48 hours, Day 7
  Measurement of body temperature in degrees Celsius at the time of the visit
Vital signs - Systolic and diastolic blood pressure | Day 0, 48 hours, Day 7
  Measurement of blood pressure in mmHg at the time of the visit
Vital signs - Heart rate | Day 0, 48 hours, Day 7
  Measurement of heart rate in beats per minute (bpm) at the time of the visit
Mortality | 3 months
  Mortality rate (%)
EQ-5D-5L | 3 months
  An instrument to describe and value health across a wide range of disease areas.
  5-level EQ-5D (EuroQol instrument with 5 dimensions and 5 levels) version with five dimensions (five levels, categorical options): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Score ranges:
  1. I have no problems ...walking/dressing, etc (better outcome);
  2. I have some problems ...walking/dressing, etc;
  3. I have moderate problems ...walking/dressing, etc;
  4. I have severe problems ...walking/dressing, etc;
  5. I have extreme problems ...walking/dressing, etc (worse outcome).
Recurrent stroke assessment | Day 0, 48 hours, Day 7
  Assessment of stroke recurrence after the first event, specifying the type into categories (no recurrence, new transient ischemic attack, new ischemic stroke, hemorrhagic stroke) and the time interval between events.
MONTREAL COGNITIVE ASSESSMENT (MoCA) | Month 3
  A brief cognitive screening tool used to assess mild cognitive impairment, score from 0-30.
  Score ranges:
  < 19: moderate to severe cognitive impairment (worse outcome); 19-25: mild cognitive impairment; > 26: normal (better outcome).
Hospital Anxiety and Depression Scale (HADS) | 3 months
  Final score of the scale that assesses anxiety and depression in patients, especially those with physical illnesses (score from 0-21, wiht 14 items and each item with four-point scale, 0-3).
  Score ranges:
  0-7: Normal - No significant symptoms of anxiety or depression (better outcome); 8-10: Borderline/Mild - Presence of symptoms that may require attention; 11 or higher: Probable Case/Severe - Clinically significan psychological disorder or "probable case" (worse outcome).
Mobility assessment | 48 hours, Day 7, Month 3.
  Assessment of participant mobility according to categories (not yet mobilized, transfers to chair, ambulating)
Breath Holding Index (BHI) - measure 1 | Before 48 hours or Day 7 (if not performed previously)
  Non-invasive method used to assess cerebrovascular reactivity, specifically the ability of the brain's blood vessels to adjust to changes in carbon dioxide levels.
  Three attempts will be performed for each participant with measurements of:
  * (a) baseline mean flow velocity before the apnea test (cm/sec)
Breath Holding Index (BHI) - measure 2 | Before 48 hours or Day 7 (if not performed previously)
  Non-invasive method used to assess cerebrovascular reactivity, specifically the ability of the brain's blood vessels to adjust to changes in carbon dioxide levels.
  Three attempts will be performed for each participant with measurements of:
  * (b) mean flow velocity at the end of the apnea test (cm/sec).
Breath Holding Index (BHI) - measure 3 | Before 48 hours or Day 7 (if not performed previously)
  Non-invasive method used to assess cerebrovascular reactivity, specifically the ability of the brain's blood vessels to adjust to changes in carbon dioxide levels.
  Three attempts will be performed for each participant with measurements of:
  * (c) apnea duration (sec).
Hemorrhagic transformation | 48 hours, Day 7
  Type of ischemic stroke complication according to hemorrhage infarction (HI) /parenchymal hemorrhage (PH) levels in brain tissue.
  Score:
  0- No complication HI1- Hemorrhage infarction 1; HI2- Hemorrhage infarction 2; PH1- Parenchymal hemorrhage 1; PH2- Parenchymal hemorrhage 2; No follow-up CT/MRI performed.
Early Mobilization Decision (<48h) | Day 0
  Ultrasound-guided (US) mobilization: early mobilization (<48h) if no cerebral hemodynamic impairment in US; Decision - yes or no? (only for interventional group)
Hospitalization duration | Month 3
  Number of days of hospitalization
White matter lesions in neuroimaging | Day 0
  White matter legions in neuroimaging - ARWMC scale: 0-no lesions (better outcome); 1-focal lesions; 2-beginning confluence of lesions; 3-diffuse involvement of the entire region, with or without involvement of U fibers (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Joao Sargento Freitas, MD, PhD, Principal Investigator — Unidade Local de Saude de Coimbra; Joao Sargento Freitas, MD, PhD, Study Director — Unidade Local de Saude de Coimbra
Locations (3):
- Portugal (3):
  - Unidade Local de Saude de Coimbra, Coimbra, Coimbra District
  - Unidade Local de Saúde de Santa Maria, Lisbon, Lisbon District
  - Unidade Local de Saúde de São João, Porto, Porto District

IPD SHARING:
Plan to Share IPD: No
Data will be irreversibly anonymized and exclusively handled by researchers involved in the study.